CLINICAL TRIAL: NCT03893136
Title: The Cohort Study of East Chinese Takayasu's Arteritis (ECTA-cohort Study)
Brief Title: The Registry Study of Takayasu Arteritis in East China
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECTA-cohort study
Record Dates: First submitted 2019-03-12; First posted 2019-03-28 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Takayasu Arteritis; Mechanisms, Defense; Pregnancy Related; Treatment Refusal; Outcome
Keywords: Takayasu arteritis; follow-up; treatment; outcome; pregnancy; cohort
MeSH Terms: conditions — Takayasu Arteritis; Treatment Refusal | interventions — tocilizumab; Leflunomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The whole blood was drawn and centrifuged to get serum, plasma, and cell pellet. The vascular specimens were also obtained with permission.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Control group: The control group mainly consists of healthy volunteers. The whole blood is obtained and frozen to detect the corresponding biochemical markers in the futures. The vascular tissues are obtained from the deserted and free abdominal aorta conjugated to the renal artery in the kidney transplantation.
- sham TA group: In the TA cohort, patients are divided into two groups mainly, sham TA group and scramble TA group. The sham TA group is the TA group who is given the traditional and classical intervention or treatment and so on.
- scramble TA group: Compared to sham TA group in the cohort, scramble TA group refers to TA patients who are given novel drugs or new drugs which are safe to treat other autoimmune diseases but have not been used to treat TA yet, or some new interventions and so on.
  Interventions: Biological: Tocilizumab; Drug: Leflunomide

INTERVENTIONS:
Biological: Tocilizumab — The scramble TA group is given bioagents such as IL-6R antibody, CD20-antibody, TNF-alpha antibody, and other bioagents which are safe to use in human to treat other refractory diseases. The sham group is given cyclophosphamide. And the prednisone is the basic drugs to be used in TA.
  Other Names: IL-6R antibody
  Groups: scramble TA group
Drug: Leflunomide — The scramble TA group is given new molecules such as Leflunomide, Iguratimod, and other molecules which are safe to use in human to treat other refractory diseases. The sham group is also given cyclophosphamide. And the prednisone is the basic drugs to be used in TA.
  Other Names: Arava
  Groups: scramble TA group

SUMMARY:
The Takayasu arteritis (TA) is a rare inflammatory large vessel arteritis which often occurs women in Aisa, one of which is China. The rare cases restricted the development of intervention strategy, especially in female patients who plan to be pregnant. So investigators try to recruit as many TA participants as possible to build a TA cohort so that investigators could manage patients much more professionally and standardized and explore the better interventional strategy for a better outcome as well, with full use of blood and vascular tissues.

DETAILED DESCRIPTION:
1. Overview of Takayasu's arteritis.

   Takayasu arteritis (TA) is a chronic inflammatory blood vessel that seriously endangers human health, which affects a large variety of blood vessels, characterized by vascular stenosis and occlusion. The clinical manifestations of TA are hypertension, renal failure caused by renal artery stenosis; pulseless, syncope and cerebral infarction caused by carotid vessels stenosis; pulmonary infarction induced by thoracic aorta involvement, etc. The TA usually accompanies high morbidity, high mortality, and poor prognosis. TA is a rare disease which is prone to occur in Asian women, especially in young women (20-40 years old) in the growth period. Currently, the etiology and pathogenesis of TA remain unclear, and the state of the disease is often repeatedly active and continuously progressive. Moreover, non-effective therapy exists for the moment.
2. The diagnosis and activity evaluation of TA

   At present, TA is diagnosed according to the American Society of Rheumatology (ACR) classification criteria for Takayasu's arteritis: ① onset at age ≤40 years; ② claudication of an extremity; ③ decreased brachial artery pulse; ④ >10 mm Hg difference in systolic blood pressure between arms; ⑤ a bruit over the subclavian arteries or the aorta; ⑥ and arteriographic evidence of narrowing or occlusion of the entire aorta, its primary branches, or large arteries in the proximal upper or lower extremities. Participants who meet 3 or more criteria could be diagnosed with this disease posterior to excluding atherosclerosis, congenital muscle fiber dysplasia, etc.

   The course of TA is often manifested as chronic, repetitive activity and continuous progression. The evaluation standard proposed by Kerr et al. to monitor TA activity is widely used clinically. Two more new emerging or aggravating clinical manifestations indicates disease Activity: ① systemic symptom, such as fever, bones, muscle symptoms; ② increased erythrocyte sedimentation rate (ESR); ③characteristics of vascular ischemia or inflammation: such as intermittent claudication, pulse weakening or pulseless, vascular bruit, vascular pain, asymmetry blood pressure, etc.; ④ abnormalities in angiography. Although acute phase response protein such as ESR and C-reactive protein (CRP) are non-specific indicators for inflammation, they are still important markers to evaluate the disease activity. Imaging follow-up, primarily based on magnetic resonance imaging (MRI) and color Doppler ultrasound, is critical in assessing TA disease activity. With the help of Pro. Jiang Lin and Dr. Lu Peng, investigators have established an imaging diagnostic team in recent years and proposed the systemic MRI scoring standard in the international firstly. The standard has been applied to quantitatively assess the vascular inflammation prior and posterior to the treatment in participants with TA. Recently, investigators co-operated with the Department of Nuclear Medicine and Radiology to employ the 18F-FDG-PET/CT to evaluate the systemic vascular inflammation and disease activity in participants. Moreover, investigators attempted to use contrast-enhanced ultrasound microbubble imaging to assess the carotid artery inflammation and stenosis. At present, these two technologies are still being explored. Therefore, it is necessary to combine the clinical manifestations, acute phase response proteins (ESR and CRP) and imaging to judge the TA disease activity comprehensively.
3. Treatment of arteritis

   The treatment of TA is divided into two phases: remission induction period and maintenance period. The drugs are divided into three categories including glucocorticoids, cytotoxic drugs, and biological agents targeting inflammatory cytokines.

   Glucocorticoids are the basic drug for TA treatment. Most TA participants receiving high doses of glucocorticoids treatment could be induced remission quickly, but about 17%-29% of refractory participants treated with standard glucocorticoids strategy could not be alleviated. And the recurrence rate is up to 90% with the single glucocorticoid. About more than 2/3 of participants would be glucocorticoid-dependent, and more than half of the participants need other drugs to maintain remission. Moreover, long-term high-dose glucocorticoids also have many adverse effects.

   Recently, targeted biological agents have been attempted to treat refractory, recurrent TA and glucocorticoid-dependent remission induction TA participants. Compared with conventional drugs, targeted biological agents work faster and could bring disease remissions for 70%-90% of refractory participants. However, the long-term use of biological agents would threaten the low-immunity participants with the risk of infections and cancer. Moreover, the effect on the reproductive system is unclear for the moment; in addition, these drugs are expensive and mainly used in refractory and critically ill participants.

   The combination of glucocorticoids combining with immunosuppressive agents such as cyclophosphamide, methotrexate, azathioprine, mycophenolate mofetil, etc. are the commonly used remission induction strategy clinically. However, large amounts of clinical evidence demonstrate that TA participants receiving glucocorticoids with the immunosuppressive agents would also face the histopathological activities lesions in the future. In the long-term follow-up, the relapse rate is much higher, and the mortality rate is significantly higher than that of healthy people.

   In summary, the current commonly used drugs for TA treatment could not meet the needs of the clinical setting, and TA participants lack a universally effective treatment strategy.
4. Pregnancy of TA participants

TA often occurs in women of childbearing age, so reducing the risk of maternal pregnancy caused by pregnancy in TA participants is one of the investigators' focuses in recent years. At present, there are no relevant guidelines for the pregnancy of TA participants, and doctors instruct them to take pills and monitor disease activity mainly basing on the doctor's clinical experience. Usually, investigators do not recommend the TA participants in active phase to conceive, not only because that the use of hormones and cytotoxic drugs could influence the development of the fetus, but also because that the stenosis or occlusion of the distal artery would increase the cardiac load so as to cause congestive heart failure, pre-eclampsia as well as fetal growth restriction and stillbirth. A case-control study in Brazil recruiting 89 TA and 89 healthy pregnant women discovered that the risk of gestational hypertension and low birth weight was much higher in TA than that in healthy controls. Moreover, the perinatal mortality rate is much higher in TA pregnant participants as well. A retrospective study in France including 96 TA pregnant women, 240 cases of pregnancy events, revealed that TA did not affect the pregnancy outcomes, but increased the risk of complications such as pregnancy hypertension with the elevating of the disease activity. Therefore, there is a lack of large-scale evidence-based medical proof uncovering the relationship between the pregnancy outcome and maternal risk in participants of TA. Here, the present follow-up registration also extends to the service of pregnant TA participants, which is designed to guide the treatment of pregnant participants and monitor maternal safety.

This objective of this study is to record the related materials of the follow-up of TA participants and the pregnancy course, to direct the standardized medication, to monitor the changes of disease conditions, and to provide the better prognosis and pregnancy outcome for TA participants.

ELIGIBILITY:
Inclusion Criteria

* onset at age ≤40 years;
* claudication of an extremity;
* decreased brachial artery pulse;
* >10 mm Hg difference in systolic blood pressure between arms;
* a bruit over the subclavian arteries or the aorta;
* angiographic evidence of narrowing or occlusion of the entire aorta, its primary branches, or large arteries in the proximal upper or lower extremities.

  * Patients should meet at least 3 of the above 6 articles.
  * Sign the informed consent

Exclusion Criteria

* autoimmune diseases, such as ANCA-associated vasculitis, systemic lupus erythematosus, Behcet's disease, rheumatoid arthritis, ankylosing spondylitis, etc.;
* complicated medical abnormal conditions, un-related with TA but engendering the unpredictable risks, such as severe, progressive, or uncontrollable kidney, liver, blood, gastrointestinal, pulmonary, heart, neuron or others
* malignant tumors;
* serious acute or chronic infections;
* high risk of tuberculosis infection such as clinical, radiological or laboratory evidence of active or occult tuberculosis, or the history of active tuberculosis;
* Having received or plan to receive plasma exchange or lymphocyte replacement or immunoabsorption therapy within 1 year.
* Preparing to receive an attenuated vaccine during the trial;
* Having received or plan to receive an organ transplant;

Exit criteria

* participants require to withdraw during the study;
* participants who believe that they need to withdraw due to clinical adverse events;
* Participants can not or does not comply with the requirements of the research protocol;

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population of the present investigation is TA patients mainly deriving from east China. The subjects are mainly female at the pregnancy age, who have the necessity to be pregnant. But there is not any drug or other intervention to cure them thoroughly.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The change of manifestations of systemic symptom - fever | Through study completion, an average of 2 months.
  The change of manifestations of systemic symptoms could effectively reflect the disease status of patients. The systemic symptoms associated with Takayasu arteritis mainly consist of fever, fatigue and chest congestion. Fever is examined by thermometer with the axillary's temperature, and the T>37.5 degree is considered to be fever. After investigators excluding the fever caused by infection through CT or laboratory examinations, the occurrence of fever usually indicates the disease activity.
The change of manifestations of systemic symptom - fatigue | Through study completion, an average of 2 months.
  The occurrence of fatigue indicates that the disease might be in the active phase. Self reported fatigue is obtained through inquiry, recorded by investigators and classified as "WITH" and "WITHOUT".
The change of manifestations of systemic symptoms - chest congestion | Through study completion, an average of 2 months.
  The occurrence of chest congestion indicates that the heart and pulmonary might be involved and the disease might be in the active phase. Self reported chest congestion is obtained through inquiry, recorded by investigators and classified as "WITH" and "WITHOUT".
The change of the emerging signs or symptoms of ischemia | Through study completion, an average of 2 months.
  Multiple emerging signs or symptoms could sensitively reflect the extent of ischemia of artery or organs. Self-reported emerging signs or symptoms of ischemia including vascular pain, dizziness, headache, amaurosis, vision loss, blurred vision, palpitations, chest pain, abdominal pain, claudication and other symptom through inquiry are recorded by investigators and classified as "WITH" and "WITHOUT". Participants with emerging signs or symptoms of ischemia usually face aggravating TA disease.
The change of the signs or symptoms of ischemia | Through study completion, an average of 2 months.
  The vascular bruits and pulse strength are evaluated and scored from 0 to 2 (0=without bruits and pulse; 1=bruits and decreased pulse; 2= normal) by a special well-trained investigator. If the score decreases, the ischemia is exacerbated and classified as "WITH".
The change of the blood pressure | Through study completion, an average of 2 months.
  The blood pressure change is measured with sphygmomanometer by the investigators. The measure is performed three times in each visit, and the mean systolic blood pressure (SBP) and mean diastolic blood pressure (DBP) are recorded. If the pressure fluctuates over 20mmHg, the stenosis of artery may exacerbate and the disease might be in the active phase.
The change of laboratory tests. | Through study completion, an average of 2 months.
  The laboratory inflammatory markers such as erythrocyte sedimentation rate (ESR) are concise and efficient methods to monitor the change of disease status, and are examined by clinical laboratory in Zhongshan Hospital of Fudan University. Investigators record and summarize the results and evaluate the change of ESR under different treatment options.
The change of IL-6 in plasma | Through study completion, an average of 2 months.
  IL-6 plays an important role in the progression of Takayasu arteritis. The level of plasma IL-6 is detected by clinical laboratory in Zhongshan Hospital of Fudan University. Investigators record and summarize the results and evaluate the change of IL-6 under different interventions, and analyze the relationship between IL-6 and disease status.
The change of vascular imaging. | Through study completion, an average of 2 months.
  MRA and contrast-enhanced carotid ultrasound imaging are important methods to evaluate TA vascular inflammation and structural change. In the initial interview and every 3 times of follow-up, the imaging examination are carried out and the images are stored at the hospital. Two radiologists perform the independent reading and evaluation. Vascular imaging is employed to monitor the improvement of the vascular wall inflammation and vascular structures (including vessel wall thickness and vascular stenosis) during treatment. For patients with stent or other metallic foreign things in the body, PET-CT and CT are also used to examine the shape and lumen of the vessels.
The change of quality of life(QOF): SF-36 questionnaire | Through study completion, an average of 2 months.
  The change of Quality of Life (QOF) with the SF-36 questionnaire Self reported the change of quality of life. Patients complete the SF-36 quality of life assessment questionnaire. Investigators provide the guidance and training on how to complete the questionnaire but must not interfere with the patients' own choice. Investigators evaluate the change of overall quality of life of patients and score the change from 0 to 2 (0= alleviated, 1=similar, 2= worsen).

SECONDARY OUTCOMES:
The change of obstetric related examinations in childbearing women. | From the initiation of pregnancy, 1 year.
  For childbearing women who are preparing to be pregnant and being pregnant, investigators pay special attention to these participants and provide proper guidance and assistance promptly. To evaluate the change of obstetric related examinations, investigators record the results of obstetric related examinations such as height of uterus, abdominal perimeter, and collaborate with ultrasound specialist to perform the obstetric ultrasound to monitor the status of fetus. At last, investigators assess the process and scores from 0 to 4 with the help of doctors from gynecologist and obstetrician. (0= much better than normal women, 1= similar to normal women, 2= worse than normal women but without obstetrics and gynecology complications, 3= worse than normal women with obstetrics and gynecology complications, 4= abortion, death of fetus or mother.)

CONTACTS AND LOCATIONS:
Overall Officials: Lindi Jiang, PhD, Study Chair — Fudan University
Locations (1):
- Department of Rheumatology in Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Direskeneli H, Aydin SZ, Merkel PA. Disease assessment in Takayasu's arteritis. Rheumatology (Oxford). 2013 Oct;52(10):1735-6. doi: 10.1093/rheumatology/ket274. Epub 2013 Aug 16. No abstract available. PMID 23955648
- [Background] Arnaud L, Haroche J, Mathian A, Gorochov G, Amoura Z. Pathogenesis of Takayasu's arteritis: a 2011 update. Autoimmun Rev. 2011 Nov;11(1):61-7. doi: 10.1016/j.autrev.2011.08.001. Epub 2011 Aug 9. PMID 21855656
- [Background] Wen D, Du X, Ma CS. Takayasu arteritis: diagnosis, treatment and prognosis. Int Rev Immunol. 2012 Dec;31(6):462-73. doi: 10.3109/08830185.2012.740105. PMID 23215768
- [Background] Fillaus JA, Oliveto J, Cutinha A, Cannella A, Plumb TJ. Takayasu arteritis presenting as new-onset hypertension. J Clin Rheumatol. 2014 Oct;20(7):389-90. doi: 10.1097/RHU.0000000000000177. No abstract available. PMID 25275769
- [Background] Arend WP, Michel BA, Bloch DA, Hunder GG, Calabrese LH, Edworthy SM, Fauci AS, Leavitt RY, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of Takayasu arteritis. Arthritis Rheum. 1990 Aug;33(8):1129-34. doi: 10.1002/art.1780330811. PMID 1975175
- [Background] Kerr GS, Hallahan CW, Giordano J, Leavitt RY, Fauci AS, Rottem M, Hoffman GS. Takayasu arteritis. Ann Intern Med. 1994 Jun 1;120(11):919-29. doi: 10.7326/0003-4819-120-11-199406010-00004. PMID 7909656
- [Background] Jiang L, Li D, Yan F, Dai X, Li Y, Ma L. Evaluation of Takayasu arteritis activity by delayed contrast-enhanced magnetic resonance imaging. Int J Cardiol. 2012 Mar 8;155(2):262-7. doi: 10.1016/j.ijcard.2010.10.002. Epub 2010 Nov 6. PMID 21059475
- [Background] O'Connor TE, Carpenter HE, Bidari S, Waters MF, Hedna VS. Role of inflammatory markers in Takayasu arteritis disease monitoring. BMC Neurol. 2014 Mar 28;14:62. doi: 10.1186/1471-2377-14-62. PMID 24678735
- [Background] Kotter I, Henes JC, Wagner AD, Loock J, Gross WL. Does glucocorticosteroid-resistant large-vessel vasculitis (giant cell arteritis and Takayasu arteritis) exist and how can remission be achieved? A critical review of the literature. Clin Exp Rheumatol. 2012 Jan-Feb;30(1 Suppl 70):S114-29. Epub 2012 May 11. PMID 22640655
- [Background] Nakaoka Y, Higuchi K, Arita Y, Otsuki M, Yamamoto K, Hashimoto-Kataoka T, Yasui T, Ikeoka K, Ohtani T, Sakata Y, Shima Y, Kumanogoh A, Yamauchi-Takihara K, Tanaka T, Kishimoto T, Komuro I. Tocilizumab for the treatment of patients with refractory Takayasu arteritis. Int Heart J. 2013;54(6):405-11. doi: 10.1536/ihj.54.405. PMID 24309452
- [Background] Youngstein T, Peters JE, Hamdulay SS, Mewar D, Price-Forbes A, Lloyd M, Jeffery R, Kinderlerer AR, Mason JC. Serial analysis of clinical and imaging indices reveals prolonged efficacy of TNF-alpha and IL-6 receptor targeted therapies in refractory Takayasu arteritis. Clin Exp Rheumatol. 2014 May-Jun;32(3 Suppl 82):S11-8. Epub 2013 Sep 30. PMID 24093733
- [Background] Mekinian A, Comarmond C, Resche-Rigon M, Mirault T, Kahn JE, Lambert M, Sibilia J, Neel A, Cohen P, Hie M, Berthier S, Marie I, Lavigne C, Anne Vandenhende M, Muller G, Amoura Z, Devilliers H, Abad S, Hamidou M, Guillevin L, Dhote R, Godeau B, Messas E, Cacoub P, Fain O, Saadoun D; French Takayasu Network. Efficacy of Biological-Targeted Treatments in Takayasu Arteritis: Multicenter, Retrospective Study of 49 Patients. Circulation. 2015 Nov 3;132(18):1693-700. doi: 10.1161/CIRCULATIONAHA.114.014321. Epub 2015 Sep 9. PMID 26354797
- [Background] Assad AP, da Silva TF, Bonfa E, Pereira RM. Maternal and Neonatal Outcomes in 89 Patients with Takayasu Arteritis (TA): Comparison Before and After the TA Diagnosis. J Rheumatol. 2015 Oct;42(10):1861-4. doi: 10.3899/jrheum.150030. Epub 2015 Sep 1. PMID 26329335
- [Background] Comarmond C, Mirault T, Biard L, Nizard J, Lambert M, Wechsler B, Hachulla E, Chiche L, Koskas F, Gaudric J, Cluzel P, Messas E, Resche-Rigon M, Piette JC, Cacoub P, Saadoun D; French Takayasu Network. Takayasu Arteritis and Pregnancy. Arthritis Rheumatol. 2015 Dec;67(12):3262-9. doi: 10.1002/art.39335. PMID 26315109